CLINICAL TRIAL: NCT07001631
Title: Effect of EMDR for Reduction of Pain Interference in Children With Sickle Cell Disease
Acronym: RELAX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Karin Fijnvandraat, prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL86274.018.24; RELAX (Other: CCMO)
Record Dates: First submitted 2025-04-28; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-03

CONDITIONS: Sickle Cell Disease; Pain; Pain, Chronic Disease
Keywords: Pain; Pain Interference; Vaso-occlusive crisis; EMDR; PTSD
MeSH Terms: conditions — Anemia, Sickle Cell; Pain; Chronic Disease; Vaso-Occlusive Crises; Stress Disorders, Post-Traumatic | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EMDR intervention group (Active Comparator): Measurements will be done for the complete study population at inclusion (T0). Participants randomized to the intervention group will start the EMDR therapy as soon as possible. After the intake session (week 1), including case conceptualization and treatment plan, a maximum of 6 weekly EMDR sessions with a duration of 1 hour per session will be offered. In the intervention group, measurements will be done 2 weeks (T1i) and 3 months (T2i) after the end of EMDR sessions.
  Interventions: Other: Eye Movement Desensitization and Reprocessing (EMDR)
- Wait-list control group (Other): Measurements will be done for the complete study population at inclusion (T0). Participants randomized to wait-list control group will wait for 9 weeks to start the therapy. Eight weeks after inclusion (T1c) will be performed for participants in the wait-list control group, just before they receive EMDR treatment. After the intake session (week 1), including case conceptualization and treatment plan, a maximum of 6 weekly EMDR sessions with a duration of 1 hour per session will be offered. Participants of the wait-list control group are asked to complete measurements 2 weeks (T1.1c) and 3 months after the end of EMDR sessions (T2c).
  Interventions: Other: Eye Movement Desensitization and Reprocessing (EMDR)

INTERVENTIONS:
Other: Eye Movement Desensitization and Reprocessing (EMDR) — The Dutch version of the standard EMDR protocol with age-specific adaptations for children and adolescents will be used. The eight phases consist of history taking, preparation, assessment, desensitization, installation, body scan, closure, and re-evaluation. During an EMDR session, the child focuses on emotionally disturbing memories (images, thoughts, emotions, and sensations) while simultaneously focusing on an external distracting stimulus (e.g., eye movements). This process facilitates accessing and desensitizing the traumatic memory network, so information processing is enhanced, and new associations can be made between the traumatic memory and more adaptive memories and information. As a result, the traumatic memory representation will be less intense and emotionally disturbing. After the intake session (week 1), including case conceptualization and treatment plan, a maximum of 6 weekly EMDR sessions with a duration of 1 hour per session will be offered.
  Other Names: EMDR therapy; EMDR treatment

SUMMARY:
Children with sickle cell disease may experience frequent painful episodes. This, together with the traumatic experiences during a hospitalization, can lead to the development of posttraumatic stress reactions. As the stress can trigger painful episodes (pain crisis) in children with sickle cell disease, the investigators think that treating these stress symptoms can reduce the pain-related problems in their lives. Eye Movement Desensitization and Reprocessing (EMDR) is proven to be an effective trauma treatment for posttraumatic stress disorder. Research studies show that EMDR can reduce pain in adults. The investigators want to study now if EMDR effective is in reducing pain-related problems in children with sickle cell disease.

DETAILED DESCRIPTION:
Objective: The primary objective of this study is to investigate the efficacy of EMDR therapy in reducing pain interference in the lives of children with SCD. Secondary objectives are to study the efficacy of EMDR in reducing PTSD symptoms, anxiety, depressive symptoms, physical complaints (low mobility), frequency and severity of pain, use of pain medication, and number of days absent from school. Themes of pain and trauma-related memories and feasibility of EMDR therapy for this population will also be explored.

Study design: In this single-center randomized controlled trial (RCT) patients (aged 6-18 years) with SCD and clinically relevant scores on PROMIS pain interference will be randomized into an intervention group and waiting list control group. Measurements will be done for the complete study population at inclusion (T0). In the intervention group, measurements will be done 2 weeks (T1i) and 3 months (T2i) after the end of EMDR sessions. Eight weeks after inclusion (T1c) will be performed for participants in the waiting list control group just before they receive EMDR treatment, and they are asked to complete measurements, 2 weeks (T1.1c) and 3 months after the end of EMDR sessions (T2c).

Intervention: After the intake session (week 1), including case conceptualization and treatment plan, a maximum of 6 weekly EMDR sessions with a duration of 1 hour per session will be offered. The waiting list control group will wait 9 weeks before starting EMDR therapy.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of SCD
* Age between 6 and 18 years old
* Elevated pain interference scores: Reporting above the clinical cut-off T-score of 49 on PROMIS Pain Interference (parent-proxy version for children from 6-7 years and self-report version for children from 8 years).
* Having sufficient knowledge of the Dutch or English languages to complete the assessments

Exclusion Criteria:

* Undergone successful stem cell transplantation
* Pregnant adolescents
* Current unsafety that is likely to interfere with psychological therapy for example ongoing domestic violence
* Major interfering acute medical or psychiatric condition, such as psychosis, substance dependence, current severe self-harm or high risk for suicide requiring immediate treatment
* Receiving psychological (trauma) treatment by another therapist at the same time
* IQ estimated to be < 80 based on information contained in the medical history or information from educational services/school

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain interference | Tscreen, inclusion (T0), 2 weeks after end of treatment (T1i/T1.1c) or 8 weeks after inclusion (T1c), 3 months after end of treatment (T2)
  The PROMIS Short Form - Pain Interference 8a for measuring Pain Interference will be used. The PROMIS Pain Interference questionnaire assesses the pain impact on relevant aspects of one's life. This includes the extent to which pain affects social, cognitive, emotional, physical, and recreational activities. It also incorporates items probing sleep and enjoyment in life. The questionnaire assesses pain interference over the past seven days (recall period). A higher PROMIS T-score represents more pain interference. This scale ranges from 0 to 100 points. In his dissertation, Luijten reports that the general Dutch pediatric population reports a mean score of 39 points with a standard deviation of 10 points. Therefore, T-scores of 49 and above represent a (sub)clinical level of functioning. On a previous study from our group, children with severe SCD phenotype (n= 36) reported a mean score of 52.73 points (SD= 12.72), while the ones with less severe SCD phenotype (n= 54).

SECONDARY OUTCOMES:
PTSD symptoms | Tscreen, inclusion (T0), 2 weeks after end of treatment (T1i/T1.1c) or 8 weeks after inclusion (T1c), 3 months after end of treatment (T2)
  The efficacy of EMDR in reducing PTSD symptoms. The Child and Adolescent Trauma Screen (CATS) questionnaire is a screening instrument based on the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for PTSD. It measures potentially traumatic events and PTSD symptoms (PTSS). The questionnaire consists of 15 items measuring traumatic events, 20 items measuring DSM-5 PTSD symptoms, and 5 items measuring psychosocial functioning, and it is administered in approximately 15 minutes. The 4-point symptom response scales indicate the reported frequency/severity of each symptom.
  For children aged 6-7 years, using the caregiver-report version, the possible score range is 0-48, and the recommended cut-off point indicative of (sub)clinically relevant levels of symptoms is 12 points or more. For children aged 8 years and older, using the self-report version, the possible score range is 0-60, and the cut-off point is 15 points or more.
Anxiety | Inclusion (T0), 2 weeks after end of treatment (T1i/T1.1c) or 8 weeks after inclusion (T1c), 3 months after end of treatment (T2)
  The efficacy of EMDR in reducing anxiety. PROMIS Anxiety questionnaires assess fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart, dizziness). They assess anxiety over the past seven days (recall period). PROMIS T-scores are calculated per version, with higher T-scores representing greater anxiety.
Depressive symptoms | Inclusion (T0), 2 weeks after end of treatment (T1i/T1.1c) or 8 weeks after inclusion (T1c), 3 months after end of treatment (T2)
  The efficacy of EMDR in reducing depressive symptoms. PROMIS Depressive Symptoms questionnaires assess negative mood (sadness, guilt), views of self (self-criticism, worthlessness), and social cognition (loneliness, interpersonal alienation), as well as decreased positive affect and engagement (loss of interest, meaning, and purpose). Somatic symptoms (changes in appetite, sleeping patterns) are not included, which eliminates consideration of these item's confounding effects when assessing children with comorbid physical conditions. The questionnaires are universal rather than disease-specific, making scores easily comparable to the general population. They assess depressive symptoms over the past seven days (recall period). The PROMIS T-scores are calculated per version. A higher PROMIS T-score represents more depressive symptoms.
Physical complaints (low moblity) | Inclusion (T0), 2 weeks after end of treatment (T1i/T1.1c) or 8 weeks after inclusion (T1c), 3 months after end of treatment (T2)
  The efficacy of EMDR in reducing physical complaints. These questionnaires assess activities of physical mobility such as getting out of bed or a chair to activities such as running. They assess mobility over the past seven days (recall period). The PROMIS T-scores are calculated per version. A higher PROMIS T-score represents more mobility.
Pain frequency | Inclusion (T0), 2 weeks after end of treatment (T1i/T1.1c) or 8 weeks after inclusion (T1c), 3 months after end of treatment (T2)
  The efficacy of EMDR in reducing pain frequency. At T0, T1i/T1.1c, T1c and T2, participants should complete a diary and report for each day of the week if they had pain (yes/no).
Pain severity | Inclusion (T0), before and after each EMDR session, 2 weeks after end of treatment (T1i/T1.1c) or 8 weeks after inclusion (T1c), 3 months after end of treatment (T2).
  The efficacy of EMDR in reducing pain severity. At T0, T1i/T1.1c, T1c and T2, participants should complete a diary and rate, for each day of the week that they had pain, the severity of the pain on a numeric rating scale (NRS, 0 - 10, 10 indicating the highest pain). It will also be investigated before and after each EMDR session using the same NRS, and will be registered by the therapist as part of the session report.
Use of pain medication | Inclusion (T0), 2 weeks after end of treatment (T1i/T1.1c) or 8 weeks after inclusion (T1c), 3 months after end of treatment (T2).
  The efficacy of EMDR in reducing pain medication use. At T0, T1i/T1.1c, T1c and T2, participants should complete a diary and report for each day of the week any pain medication used. The (multiple-choice) options available are: no pain medication, paracetamol, diclofenac/ibuprofen, tramadol.
School absence | Inclusion (T0), 2 weeks after end of treatment (T1i/T1.1c) or 8 weeks after inclusion (T1c), 3 months after end of treatment (T2)
  The efficacy of EMDR in reducing school absence. At T0, T1i/T1.1c, T1c and T2, participants should complete a diary and report for each day of the week if they went to school (yes/no; if 'no' is chosen, they can also answer why, in a free text format).

OTHER OUTCOMES:
Feasibility of EMDR intervention | 2 weeks after end of treatment (T1i/T1.1c)
  EMDR treatment feasibility will be evaluated via a semi-structured interview performed by the researcher with the participants.
Pain and trauma related targets | Through intervention (intake and EMDR sessions), an average of 7 weeks.
  The investigators aim to describe and summarize the pain-related traumatic experiences and irrational fears of the future that exist among the children in our target group.
  During the intake, the psychologist will follow the standard procedure, in which the participant's pain-related traumatic experiences (targets) and irrational fears of the future (flash forwards) are identified by developing a case conceptualization, including a hierarchy in which these memories will be treated.
  The investigators will create a systematic description (summary of intake's data) of these identified experiences and irrational fears of the future.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Fijnvandraat, prof. dr., Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided